CLINICAL TRIAL: NCT03496311
Title: Effects of Pregnancy on the Physico-chemical Characteristics of Cerebrospinal Acid-base Equilibrium
Brief Title: Cerebrospinal Acid-base in Pregnant and Non-pregnant Fertile Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: University of Milan (Other)
Responsible Party: Sponsor
Other Study IDs: CSF acid-base in pregnancy
Record Dates: First submitted 2018-03-29; First posted 2018-04-12 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Acid-Base Imbalance; Respiratory Alkalosis; Cerebrospinal Fluid; Pregnancy
MeSH Terms: conditions — Acid-Base Imbalance; Alkalosis, Respiratory

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — samples of plasma and cerebrospinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant Women: Pregnant women with gestational age > 35 weeks undergoing spinal anesthesia for elective cesarean section.
  Interventions: Diagnostic Test: Acid - Base characterization
- Control Group: Fertile, non-pregnant women undergoing spinal anesthesia for elective surgery.
  Interventions: Diagnostic Test: Acid - Base characterization

INTERVENTIONS:
Diagnostic Test: Acid - Base characterization — Samples of cerebrospinal fluid and arterial blood will be collected anaerobically to measure acid-base variables, electrolytes, albumin, progesterone and copeptin levels

SUMMARY:
The third trimester of pregnancy is typically characterized by the development of a marked respiratory alkalosis. The possible role of pregnancy-induced variations of cerebrospinal fluid (CSF) acid-base characteristics on the development of hypocapnic alkalosis is still unknown.

Aim of this study is to characterize, according to Stewart's approach, the acid-base equilibrium of CSF and arterial plasma of pregnant women and compare the results with data obtained from fertile, non-pregnant women.

DETAILED DESCRIPTION:
The reduction in plasma PCO2 correlates with gestational age and was shown to be associated to plasma progesterone concentrations. We hypothesize that pregnancy-related haemodilution, inducing a reduction in CSF Strong Ion Difference (SID), might have a role in the development of pregnancy-related hypocapnic alkalosis.

Samples of CSF and arterial plasma of pregnant women with gestational age > 35 weeks undergoing spinal anesthesia for elective caesarean section will be analyzed for blood gases, pH, electrolytes, osmolality, albumin and haemoglobin concentration. In addition plasma copeptin levels will be analyzed. The same measurements will be performed in fertile, non-pregnant women undergoing spinal anesthesia for elective surgery.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy with gestational age > 35 weeks
* Scheduled elective cesarean section under spinal anesthesia

Exclusion Criteria:

* known respiratory or neurologic disease
* multiple pregnancies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women undergoing spinal anesthesia either for elective cesarean section of for elective surgery.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-04-13 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Strong Ion Difference | 1 day
  Strong Ion Difference (expressed in milliequivalents per Liter [mEq/L]) of cerebrospinal fluid and arterial plasma

SECONDARY OUTCOMES:
Partial pressure of carbon dioxide (PCO2) | 1 day
  PCO2 (expressed in millimeters of Mercury [mmHg]) of cerebrospinal fluid and arterial plasma
Sum of albumin (expressed in mmol/L) and Phosphates (expressed in mmol/L) | 1 day
  The total amount of weak non carbonic acids, i.e. the sum of albumin and phosphates (both expressed in mmol/L) of cerebrospinal fluid and arterial plasma
Difference between cerebrospinal fluid and arterial plasma Strong Ion Difference (Delta SID) | 1 day
  The difference between plasma and cerebrospinal fluid SID (expressed in mEq/L) will be calculated as marker of electrolyte inbalance between these two extracellular fluid compartments. Delta SID = SIDcsf - SIDplasma
Difference between cerebrospinal fluid and arterial plasma partial pressure of CO2 (Delta PCO2) | 1 day
  The difference between cerebrospinal fluid and arterial plasma PCO2 (expressed in mmHg) will be calculated as a marker of acid-base equilibrium between these two extracellular fluid compartments. Delta PCO2 = SIDplasma - SIDcsf
Progesterone levels | 1 day
  Plasma and CSF Progesterone levels (expressed in ng/mL) will be measured
Copeptin levels | 1 day
  Plasma copeptin levels (expressed in pmol/L) will be measured as a marker of antidiuretic hormone activity

OTHER OUTCOMES:
SID PCO2 correlation | 1 day
  Correlation between CSF SID and PCO2
Osmolality PCO2 correlation | 1 day
  Correlation between CSF osmolality and PCO2
Plasma progesterone PCO2 correlation | 1 day
  Correlation between plasma progesterone concentration and plasma PCO2
CSF progesterone PCO2 correlation | 1 day
  Correlation between CSF progesterone concentration and CSF PCO2

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Langer, MD, Principal Investigator — University of Milan; Antonio Pesenti, MD, Study Director — University of Milan; Edoardo Calderini, MD, Study Chair — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico di Milano; Giorgio Giudici, MD, Study Chair — University of Milan; Mariateresa Ambrosini, MD, Study Chair — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico di Milano
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy

REFERENCES:
- [Derived] Zadek F, Giudici G, Ferraris Fusarini C, Ambrosini MT, di Modugno A, Scaravilli V, Zanella A, Fumagalli R, Stocchetti N, Calderini E, Langer T. Cerebrospinal fluid and arterial acid-base equilibria in spontaneously breathing third-trimester pregnant women. Br J Anaesth. 2022 Nov;129(5):726-733. doi: 10.1016/j.bja.2022.07.048. Epub 2022 Sep 10. PMID 36096944